CLINICAL TRIAL: NCT05607394
Title: Prevalence of Tick-borne Encephalitis (TBE) in the Pediatric Population Treated at the University Hospitals of Strasbourg (HUS) and Characterization of Confirmed Pediatric Cases
Brief Title: Prevalence of Tick-borne Encephalitis in the Pediatric Population Treated at the HUS and Characterization of Confirmed Pediatric Cases
Acronym: TBE-KID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8725
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Tick-borne Encephalitis
Keywords: Tick-borne encephalitis (TBE); Genus Ixodes; TBEV infection; TBEV infection in children; Prevalence of TBE
MeSH Terms: conditions — Encephalitis, Tick-Borne

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tick-borne encephalitis (TBE) is a zoonosis mainly transmitted to humans by the bite of ticks of the genus Ixodes and, to a lesser extent, by the consumption of contaminated and unpasteurized dairy products. During the last decade, the epidemiology of this arbovirosis has changed profoundly with the discovery of new human cases and/or new areas of circulation of tick-borne encephalitis virus (TBEV) throughout Europe and particularly in France. Historically, Alsace is the main endemic area for this pathology in France. The pathology is notifiable since June 2021 in France.

Although TBEV infection in children seems to lead to a milder clinical presentation, data are much less abundant than in adults and only a few cases reported in infants under 1 year old have been published. Data from the most recent ECDC Annual Epidemiological Report on TBE (2019) showed incidence rates of approximately 0.2 and 0.5 per 100,000 population in patients younger than 5 and 15 years, respectively.

However, several observations may moderate and challenge both the low incidence rate and the less severe clinical presentation reported in children

ELIGIBILITY:
Inclusion criteria:

* Minor subject (≤ 16 years)
* hospitalized at the University Hospital of Strasbourg between 01/01/2020 and 31/12/2022
* having had a CSF sample taken as part of care, without infectious (other than TBE) or non-infectious etiology diagnosed
* whose parental authority holders have already given their consent for their child's biological resources to be kept in the "Microbiology" biocollection and reused for scientific research purposes.

Exclusion criteria:

* Patient or parental authority holders who have expressed their opposition to participate in the study
* Any person, male or female, over 16 years of age,
* or any person, male or female, under 16 years of age, treated at the University Hospitals of Strasbourg from January 2020 to December 2022, who has had a CSF sample taken as part of their care, for which a non-infectious etiology or an infectious etiology other than TBE has been diagnosed.
* Impossible to give the subject informed information (difficulties in understanding the subject, ...)

Ages: 0 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Minor subject (≤ 16 years) having had a CSF sample taken as part of care, without infectious (other than TBE) or non-infectious etiology diagnosed.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-08-24 (Estimated); Study Completion 2023-10-24 (Estimated)

PRIMARY OUTCOMES:
Determining the prevalence of TBE in pediatric patients (aged 0 to 15 years) | 2 years after infection with tick-borne encephalitis (TBE)

CONTACTS AND LOCATIONS:
Locations (1):
- Service Laboratoire de Virologie - PTM - CHU de Strasbourg - France, Strasbourg, France